CLINICAL TRIAL: NCT02249091
Title: An Investigator-Initiated Study To Evaluate Ara-C and Idarubicin in Combination With the Selective Inhibitor Of Nuclear Export (SINE) Selinexor (KPT-330) in Patients With Relapsed Or Refractory AML
Brief Title: A Phase II Study of Selinexor Plus Cytarabine and Idarubicin in Patients With Relapsed/Refractory Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GSO Global Clinical Research BV (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SAIL; 2014-000526-37 (EudraCT Number)
Record Dates: First submitted 2014-09-16; First posted 2014-09-25 (Estimated); Results first posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Acute Myeloid Leukemia (Relapsed/Refractory)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — selinexor; Idarubicin; Cytarabine

STUDY DESIGN:
Intervention Model Description: In the initial protocol, 25 patients are included in the clinical trial on the schedule described as cohort 1. After an amendment 15 further patients are included on the schedule described as cohort 2.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 / Selinexor 40 mg/m^2 in combination with cytarabine and idarubicin (Experimental): All enrolled patients are treated with cytarabine at a dose of 100 mg/m² continuous infusion (day 1-7) and idarubicin at a dose of 10 mg/m^2 iv (day 1,3,5) every 4 weeks and selinexor for up to 2 induction cycles. If a second cycle is applied idarubicin is only given on day 1 and 3.
  Selinexor is administered at a dose of 40 mg/m^2 twice weekly orally starting on day 2 (total of 8 doses per induction cycle).
  Interventions: Drug: Selinexor; Drug: Idarubicin; Drug: Cytarabine
- Cohort 2 / Selinexor 60 mg flat dose in combination with cytarabine and idarubicin (Experimental): All enrolled patients are treated with cytarabine at a dose of 100 mg/m^2 continuous infusion (day 1-7) and idarubicin at a dose of 10 mg/m^2 iv (day 1,3,5) every 4 weeks and selinexor for up to 2 induction cycles. If a second cycle is applied idarubicin is only given on day 1 and 3.
  Selinexor is administered at a flat dose of 60 mg twice weekly orally in weeks 1-3 of a 4-week cycle starting on day 2 (total of 6 doses per induction cycle).
  Interventions: Drug: Selinexor; Drug: Idarubicin; Drug: Cytarabine

INTERVENTIONS:
Drug: Selinexor — Patients receive Selinexor as specified in arm/group description (8 doses of 40 mg/m^2 or 6 doses of 60 mg per induction cycle).
  Other Names: KPT-330
Drug: Idarubicin — Infusion, iv, 10 mg/m^2, on days 1,3,5 in cycle 1, on days 1,3 in cycle 2
Drug: Cytarabine — Continuous infusion day 1 to 7, 100 mg/m^2, iv,
  Other Names: Ara-C

SUMMARY:
Acute Myeloid Leukemia (AML) is currently treated with chemotherapy by combining several drugs with different ways of inhibiting the cell growth. In this trial, standard chemotherapeutics that have proven their effectiveness for years, Ara-C and Idarubicin, will be combined with a new drug called Selinexor.

Selinexor inhibits the growth of cancer cells by keeping certain proteins in the nucleus which control the cell growth.

ELIGIBILITY:
Inclusion Criteria:

1. Cytological or histological diagnosis of AML with the exception of promyelocytic leukemia (AML M3)
2. Patients must have relapsed/refractory disease (relapse after stem cell transplantation is permitted) as defined as:

   1. patients with <PR after first cycle of induction chemotherapy, or
   2. patients with <CR(i) after second cycle of induction chemotherapy, or
   3. patients who relapse after conventional chemotherapy or
   4. patients who have undergone a single stem cell transplantation and who have relapse of their AML.
3. Men and women aged ≥18 years and eligible for standard dose of chemotherapy (7+3);
4. A period of at least 3 weeks needs to have elapsed since last treatment (with the exception of hydroxyurea) before participating in this study. Hydroxyurea induction therapy to reduce peripheral blast counts is permitted prior to initiation of treatment on protocol. Treatment may begin in <3 weeks from last treatment if deemed in the best interest of the patient after discussion with the PI of the study;
5. ECOG performance status ≤ 2
6. Serum biochemical values with the following limits unless considered due to leukemia: creatinine ≤2 mg/dl; total bilirubin ≤2x ULN, unless increase is due to hemolysis or congenital disorder; transaminases (SGPT or SGOT) ≤2.5x ULN.
7. Ability to swallow and retain oral medication;
8. Ability to understand and provide signed informed consent;
9. Cardiac ejection fraction must be >/=50% (by echocardiography).
10. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Treatment with any investigational agent within four weeks.
2. Cumulative anthracycline dose (daunorubicin or equivalent) >360 mg/m^2
3. HIV infection
4. Presence of any medical or psychiatric condition which may limit full compliance with the study, including but not limited to:
5. Presence of CNS leukemia
6. Unresolved toxicity from previous anti-cancer therapy or incomplete recovery from surgery.
7. For patients after SCT as part of prior treatment:

   1. Necessity of immunosuppressive drugs
   2. GvHD > grade 1
8. Any of the following within the 12 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis, or other thromboembolic event.
9. Ongoing cardiac dysrhythmias of NCI CTCAE >/= Grade 2.
10. Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.
11. Clinically significant bleeding within 1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-09; Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 43 patients were registered in the clinical trial at 3 sites. One patient was a screening failure. Of the remaining 42 patients, the first 27 patients were treated in cohort 1 (Selinexor dosed by Body Surface Area [BSA] 40 mg/m^2 per dose) and the other 15 patients were treated in cohort 2 (flat dose of Selinexor of 60 mg per dose).
Groups:
- Cohort 1 / Selinexor 40 mg/m^2 in Combination With Cytarabine and Idarubicin: Induction cycle: All enrolled patients were treated with selinexor, cytarabine and idarubicin as follows:
  Selinexor: 40 mg/m^2 twice weekly orally starting on day 2 (total of 8 doses per 4-week induction cycle).
  Idarubcin: i.v. infusion, 10 mg/m^2, on days 1,3,5 in cycle 1
  Cytarabine: continuous i.v. infusion day 1-7, 100 mg/m^2
  Up to two induction cycles were administered. If a second cycle was applied idarubicin was only given on days 1 and 3.
- Cohort 2 / Selinexor 60 mg Flat Dose in Combination With Cytarabine and Idarubicin: Induction cycle: All enrolled patients were treated with selinexor, cytarabine and idarubicin as follows:
  Selinexor: 60 mg flat dose twice weekly orally during weeks 1-3 of a 4-week cycle (day 2, 4, 9, 11, 16, 18; total of 6 doses per 4-week induction cycle).
  Idarubcin: i.v. infusion, 10 mg/m^2, on days 1,3,5 in cycle 1.
  Cytarabine: continuous i.v. infusion day 1-7, 100 mg/m^2
  Up to two induction cycles were administered. If a second cycle was applied idarubicin was only given on days 1 and 3.
Period: Overall Study
Arm/Group | Cohort 1 / Selinexor 40 mg/m^2 in Combination With Cytarabine and Idarubicin | Cohort 2 / Selinexor 60 mg Flat Dose in Combination With Cytarabine and Idarubicin
Started | 27 | 15
Completed | 7 | 2
Not Completed | 20 | 13
Not completed — Lack of Efficacy | 8 | 3
Not completed — Physician Decision | 4 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Death | 3 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Stable disease with following SCT | 0 | 1
Not completed — Ongoing bone marrow aplasia, periph. pancytopenia | 0 | 1
Not completed — CR with subsequent donor lymphocyte infusion | 1 | 0
Not completed — Refractory AML | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 / Selinexor 40 mg/m^2 in Combination With Cytarabine and Idarubicin | Cohort 2 / Selinexor 60 mg Flat Dose in Combination With Cytarabine and Idarubicin | Total
Number analyzed (Participants) | 27 | 15 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (15.18) | 58.5 (13.55) | 55.6 (14.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 16 | 9 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 27 | 14 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 27 | 15 | 42
Leukemia diagnosis [Count of Participants; unit: Participants]
  De Novo Acute Myeloid Leukemia (AML) | 19 | 12 | 31
  Therapy-induced AML | 2 | 0 | 2
  Secondary AML | 6 | 3 | 9
Prior stem cell transplantation (SCT) [Count of Participants; unit: Participants] | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With CR/CRi = Overall Reponse Rate
Description: Efficacy of selinexor in combination with standard chemotherapy in patients with relapsed/refractory AML by determination of rate of complete response (CR) or morphologic complete response with incomplete blood count recovery (CRi), as defined by the recommendations on diagnosis and management of AML in adults from an international expert panel, on behalf of the European LeukemiaNet:
  CR: Absolute Neutrophil count (ANC) >1.0x10^9/L, Platelet count >100x10^9/L, Bone marrow blasts <5%, no Auer rods, no evidence of extramedullary disease.
  CRi: Same as CR, but ANC may be <1.0x10^9/L and/or Platelet count <100x10^9/L.
  Patients with morphologic leukemia free-state (MLFS) were included in the group of responders. MLFS: Bone marrow blasts <5%, no Auer rods, no evidence of extramedullary disease.
  The best response after Selinexor treatment was analyzed, thus the best response after the induction cycle(s).
Time Frame: 1-2 induction cycles (4 - 8 weeks)
Population: All patients who have received study medication at least once and for whom post-baseline efficacy data upon treatment was available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 / Selinexor 40 mg/m^2 in Combination With Cytarabine and Idarubicin | Cohort 2 / Selinexor 60 mg Flat Dose in Combination With Cytarabine and Idarubicin
Number analyzed (Participants) | 27 | 15
Participants | 15 | 6

2. Secondary Outcome: Number of Participants With Partial Remission (PR) = Rate of PR
Description: Efficacy of selinexor in combination with standard chemotherapy in patients with relapsed/refractory AML by determination of rate of partial remission(PR) as defined by the recommendations on diagnosis and management of AML in adults from an international expert panel, on behalf of the European LeukemiaNet:
  PR: Absolute Neutrophil count (ANC) >1.0x10^9/L, Platelet count >100x10^9/L, at least a 50% decrease in the percentage of marrow aspirate blasts to 5-25%, or marrow blasts <5% with persistent Auer rods.
  The best response after Selinexor treatment was analyzed, thus the best response after the induction cycle(s).
Time Frame: 1-2 induction cycles (4 - 8 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 / Selinexor 40 mg/m^2 in Combination With Cytarabine and Idarubicin | Cohort 2 / Selinexor 60 mg Flat Dose in Combination With Cytarabine and Idarubicin
Number analyzed (Participants) | 27 | 15
Participants | 0 | 0

3. Secondary Outcome: Percentage of Patients Transplanted After Induction Therapy (Stem Cell Transplantation)
Description: Percentage of patients being transplanted after induction therapy (stem cell transplantation)
Time Frame: 1-2 induction cycles (4 - 8 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 / Selinexor 40 mg/m^2 in Combination With Cytarabine and Idarubicin | Cohort 2 / Selinexor 60 mg Flat Dose in Combination With Cytarabine and Idarubicin
Number analyzed (Participants) | 27 | 15
Participants | 11 | 4

4. Secondary Outcome: Early Death Rate
Description: Early death was defined as death before the end of the first induction cycle.
Time Frame: 1 induction cycle (4 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 / Selinexor 40 mg/m^2 in Combination With Cytarabine and Idarubicin | Cohort 2 / Selinexor 60 mg Flat Dose in Combination With Cytarabine and Idarubicin
Number analyzed (Participants) | 27 | 15
Participants | 0 | 4

5. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was calculated from the date of informed consent to the date of death. Patients still alive at the end of follow-up were censored at the last date of follow-up.
Time Frame: Time from registration to event, max 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 / Selinexor 40 mg/m^2 in Combination With Cytarabine and Idarubicin | Cohort 2 / Selinexor 60 mg Flat Dose in Combination With Cytarabine and Idarubicin
Number analyzed (Participants) | 27 | 15
months | 12.6 [4.2 to NA] — Not available due to low number of events | 8.0 [0.89 to NA] — Not available due to low number of events

6. Secondary Outcome: Relapse-Free Survival
Description: Relapse-free survival (RFS) was calculated from the date of CR/CRi until death or relapse, whichever occurred first. Patients were censored on the date of the last follow-up if they were alive without relapse.
Time Frame: Time from registration to event, max 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 / Selinexor 40 mg/m^2 in Combination With Cytarabine and Idarubicin | Cohort 2 / Selinexor 60 mg Flat Dose in Combination With Cytarabine and Idarubicin
Number analyzed (Participants) | 15 | 6
months | 10.9 [2.8 to NA] — Not available due to low number of events | NA [4.1 to NA] — Not available due to low number of events

7. Secondary Outcome: Event-Free Survival
Description: Event-free survival (EFS) was calculated from the time of informed consent until death, not achieving CR/CRi or relapse after CR/CRi.
Time Frame: Time from registration to event, max 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 / Selinexor 40 mg/m^2 in Combination With Cytarabine and Idarubicin | Cohort 2 / Selinexor 60 mg Flat Dose in Combination With Cytarabine and Idarubicin
Number analyzed (Participants) | 27 | 15
months | 5.6 [2.9 to 12.6] | 4.3 [0.9 to 10.4]

8. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival (PFS) was calculated from the time of informed consent to the date of recurrence or death, whichever occurred first. Patients were censored at the date of the last follow-up visit if they were alive without relapse.
  Disease progression was defined as presence of >50% increase in bone marrow blasts to a level of at least 50% and/or a doubling of the percentage of peripheral blood blasts to a level of at least 50%.
Time Frame: Time from registration to event, max 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 / Selinexor 40 mg/m^2 in Combination With Cytarabine and Idarubicin | Cohort 2 / Selinexor 60 mg Flat Dose in Combination With Cytarabine and Idarubicin
Number analyzed (Participants) | 27 | 15
months | 6.3 [2.3 to 26.3] | 4.3 [0.9 to 12.9]

ADVERSE EVENTS:
Time Frame: Throughout the treatment period from start of treatment until one month after the last dose of study mediation, on average 2 months.
Description: All patients taking at least one dose of study medication were included in the safety population. This applied to all 42 patients included.
Arm/Group | Cohort 1 / Selinexor 40 mg/m^2 in Combination With Cytarabine and Idarubicin | Cohort 2 / Selinexor 60 mg Flat Dose in Combination With Cytarabine and Idarubicin
All-Cause Mortality (participants affected / at risk) | 16/27 | 9/15
Serious Adverse Events (participants affected / at risk) | 12/27 | 8/15
Other Adverse Events (participants affected / at risk) | 27/27 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 / Selinexor 40 mg/m^2 in Combination With Cytarabine and Idarubicin (N=27) | Cohort 2 / Selinexor 60 mg Flat Dose in Combination With Cytarabine and Idarubicin (N=15)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 (0) | 2 (2) — Bone marrow aplasia
Asystole (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
General weakness (General disorders) | 1 (1) | 0 (0)
SIRS (General disorders) | 1 (1) | 0 (0) — Systemic inflammatory response syndrome
GvHD (Immune system disorders) | 1 (1) | 0 (0) — Graft-versus-host-disease
Hemophagocytosis syndrome (Immune system disorders) | 0 (0) | 1 (1) — Lymphohistiocytic syndrome, assessed as related to selinexor; cause of patient's death according to autopsy report: hemophagocytosis syndrome with acute cardiac decompensation
Lung infection (Infections and infestations) | 3 (3) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) — Neutropenia
Stroke (Nervous system disorders) | 1 (1) | 0 (0) — Reported as Multiple Brain Infarctions
Subarachnoidal hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 / Selinexor 40 mg/m^2 in Combination With Cytarabine and Idarubicin (N=27) | Cohort 2 / Selinexor 60 mg Flat Dose in Combination With Cytarabine and Idarubicin (N=15)
Nausea (Gastrointestinal disorders) | 23 (49) | 13 (19)
Diarrhea (Gastrointestinal disorders) | 24 (99) | 11 (32)
Vomiting (Gastrointestinal disorders) | 22 (46) | 9 (13)
Anorexia (Metabolism and nutrition disorders) | 22 (40) | 8 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 23 (30) | 5 (27)
Fatigue (General disorders) | 18 (23) | 9 (15)
White blood cell decreased (Investigations) | 17 (21) | 9 (23)
Platelet count decreased (Investigations) | 19 (33) | 7 (23)
Anemia (Blood and lymphatic system disorders) | 20 (33) | 5 (27)
Hypokalemia (Metabolism and nutrition disorders) | 17 (27) | 2 (2)
Hypotension (Vascular disorders) | 12 (16) | 7 (7)
Neutrophil count decreased (Investigations) | 12 (14) | 6 (15)
Mucositis oral (Gastrointestinal disorders) | 12 (19) | 6 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 8 (13)
Dizziness (Nervous system disorders) | 9 (12) | 6 (6)
Constipation (Gastrointestinal disorders) | 7 (8) | 7 (10)
Injection site reaction (General disorders) | 10 (12) | 3 (5)
Lung infection (Infections and infestations) | 8 (13) | 4 (7)
Edema limbs (General disorders) | 6 (8) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 10 (10) | 1 (1)
Sepsis (Infections and infestations) | 7 (7) | 3 (4)
Depression (Psychiatric disorders) | 5 (5) | 3 (3)
Headache (Nervous system disorders) | 5 (10) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4) | 4 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Hematoma (Vascular disorders) | 5 (7) | 2 (3)
Insomnia (Psychiatric disorders) | 5 (6) | 2 (2)
Fever (General disorders) | 2 (2) | 5 (9)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 3 (4)
Syncope (Nervous system disorders) | 5 (5) | 1 (1)
Creatinine increased (Investigations) | 3 (3) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (5) | 1 (1)
Catheter related infection (Infections and infestations) | 4 (4) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (6) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (6) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 3 (4) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 4 (4) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Toothache (Gastrointestinal disorders) | 4 (5) | 0 (0)
Allergic reaction (Immune system disorders) | 2 (3) | 2 (2)
Weight loss (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 2 (2) | 1 (1)
Blurred vision (Eye disorders) | 3 (3) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 3 (4) | 0 (0)
Edema face (General disorders) | 3 (3) | 0 (0)
Sinusitis (Infections and infestations) | 3 (4) | 0 (0)
Weight gain (Investigations) | 2 (2) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (3) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT02249091/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT02249091/SAP_001.pdf